CLINICAL TRIAL: NCT06702891
Title: Integrative Analysis of Exosome-Mediated Single-Cell Transcriptomics and Proteomics in Gastric Cardia Cancer
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024SDU-QILU-2
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cardia Cancer
Keywords: Gastric Cardia Cancer; Single-Cell RNA Sequencing; Exosomes; Proteomics
MeSH Terms: interventions — Single-Cell Gene Expression Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case group: The case group includes high-grade intraepithelial neoplasia of the stomach, early gastric cancer, and advanced gastric cancer.
  Interventions: Other: Detection of biological samples based on exosome sequencing, proteomics and single-cell RNA sequencing
- control group: Pathological findings in the control group showed no malignant changes in the stomach, including normal gastric mucosa, superficial gastritis, non atrophic gastritis, and gastric polyps, etc.
  Interventions: Other: Detection of biological samples based on exosome sequencing, proteomics and single-cell RNA sequencing

INTERVENTIONS:
Other: Detection of biological samples based on exosome sequencing, proteomics and single-cell RNA sequencing — The researchers combined exosome sequencing, proteomics and single-cell RNA sequencing to explore the heterogeneity of cardia cancer, identify specific biomarkers and potential therapeutic targets for cardia cancer.

SUMMARY:
This is an observational study with a case control design. This study included patients with gastric cancer confirmed by pathological diagnosis of gastric tissue, and matched the control population according to age, gender, etc. In this study, researchers collected clinical information and multiple biological samples such as serum and tissue tissue from the study subjects. The researchers combined exosome sequencing, proteomics and single-cell RNA sequencing to explore the heterogeneity of cardia cancer, identify specific biomarkers and potential therapeutic targets for cardia cancer, and provide a basis for the development of new diagnostic tools and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Study population signing informed consent form
* Age: 18 years old or older
* The study population must underwent endoscopic examination and was confirmed by pathological diagnosis as gastric cancer: including high-level intraepithelial neoplasia, early gastric cancer, and advanced gastric cancer.

Exclusion Criteria:

* Those who have undergone gastrointestinal surgery within the past 1 year; Patients who have undergone neoadjuvant chemotherapy and have developed tumors in the residual stomach after previous partial gastrectomy.
* Those who have used proton pump inhibitors, antibiotics, probiotics, and prebiotics daily within the past month, and those who have recently received hormone therapy.
* People with infectious diseases and other digestive system diseases that interfere with the experimental results, such as inflammatory bowel disease, irritable bowel syndrome, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case:
  The population in the case group signed an informed consent form, aged 18 years old or older. All subjects underwent endoscopic examination and were confirmed by pathological diagnosis as gastric cancer, including high-grade intraepithelial neoplasia, early gastric cancer, and advanced gastric cancer.
  Control:
  The age and gender of the study subjects in the control group were matched to the study population in the case group. The pathological results of the stomach of all subjects showed no malignant changes, including normal gastric mucosa, superficial gastritis, non atrophic gastritis, and gastric polyps, etc.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Differential protein | 6 months

SECONDARY OUTCOMES:
Key miRNA | 10 months
Differential cell subsets | 12 months
  Differential cell subsets between cardiac cancer tissue and normal tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China